CLINICAL TRIAL: NCT01194128
Title: Intervention to Facilitate Family Caregiver Adaptation to Nursing Home Transition
Brief Title: Facilitating Caregiver Adaptation to Patient Institutionalization
Acronym: FACTS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Richard Schulz, Prof. of Psychiatry, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R01NR009573 (NIH)
Record Dates: First submitted 2010-09-01; First posted 2010-09-02 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Dementia; Stroke; Heart Disease
Keywords: caregivers,; institutionalization,; dementia patients,; bereavement,; grief; complicated grief
MeSH Terms: conditions — Dementia; Stroke; Heart Diseases

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Psychoeducatioinal Support (Experimental): The intervention is comprised of three modules (see Table 6), each of which has multiple components. Module One provides basic education about the clinical aspects of frailty as well as the organization and operating procedures of long-term care facilities. Module Two focuses on advanced care planning, and Module Three is designed to improve the emotional well-being of family caregivers. The intervention will be delivered via 11 sessions lasting approximately 90 minutes each distributed over a six-month period. All family caregivers will begin with the Basic Knowledge Module. Modules Two and Three will be delivered in alternating sessions, based on caregiver need and preference, a strategy successfully used in the REACH intervention trial.
  Interventions: Behavioral: Psychoeducational Support
- INformation only control group (Active Comparator): Participants in the control group will receive a portion of the standardized packet of written information that is also provided to the treatment group. This packet will contain several fact sheets from a nationally-recognized expert source in caregiving (the Family Caregiver Alliance's National Center on Caregiving) and a national information and advocacy group (the National Citizens' Coalition for Nursing Home Reform). The fact sheets are relevant to the placement of a family member into a nursing home and are linked to the content areas covered in the intervention. Documents in this packet include "Caregiving and Depression," "End of Life Decision Making," and "Taking Care of You: Self-Care for Family Caregivers" from the Family Caregiver Alliance; and "Family Involvement in Nursing Home Care," "Problem Solving," and "Residents' Rights" from the National Citizen's Coalition.
  Interventions: Behavioral: Information only control group

INTERVENTIONS:
Behavioral: Psychoeducational Support — The intervention is comprised of three modules, each of which has multiple components. Module One provides basic education about the clinical aspects of frailty as well as the organization and operating procedures of long-term care facilities. Module Two focuses on advanced care planning, and Module Three is designed to improve the emotional well-being of family caregivers. The intervention will be delivered via 11 sessions lasting approximately 90 minutes each distributed over a six-month period. All family caregivers will begin with the Basic Knowledge Module. Modules Two and Three will be delivered in alternating sessions, based on caregiver need and preference, a strategy successfully used in the REACH intervention trial.
  Arms: Psychoeducatioinal Support
Behavioral: Information only control group — Participants in the control group will receive a portion of the standardized packet of written information that is also provided to the treatment group. The fact sheets are relevant to the placement of a family member into a nursing home and are linked to the content areas covered in the intervention. Documents in this packet include "Caregiving and Depression," "End of Life Decision Making," and "Taking Care of You: Self-Care for Family Caregivers" from the Family Caregiver Alliance; and "Family Involvement in Nursing Home Care," "Problem Solving," and "Residents' Rights" from the National Citizen's Coalition. Also provided will be a resource guide containing local contact information.
  Arms: INformation only control group

SUMMARY:
This study will assess the effects of an intervention targeting family caregivers who recently placed a relative in a long-term care facility because of cognitive and/or physical disability. In a two group randomized clinical trial we predict that caregivers assigned to active treatment will have lower levels of depressive symptoms, anxiety symptoms, and greater satisfaction with the long-term care facility when compared to individuals assigned to the control condition.

DETAILED DESCRIPTION:
This study is designed to address three interrelated needs of caregivers who recently placed a relative in a long-term care facility: (a) psychiatric problems, particularly depression and anxiety which are common among caregivers who recently placed their relative; (b) knowledge about the nature of long-care procedures and resident trajectories; and (c) end-of-life planning for the institutionalized relative. These needs will be addressed with an intervention that has three components: (a) a treatment protocol for depressive symptoms, major depression, and anxiety; (b) education about the organization and operating procedures of long-term care facilities, the clinical aspects of frailty, and a negotiated plan for caregiver participation in the care of their relative; and (c) education about resident trajectories in long-term care and assistance with end-of life planning. Expected outcomes include reduced depression and anxiety, greater satisfaction with the long-term care facility, and reduced service use because of an articulated end-of-life plan. Because this intervention is designed to reduce distress prior to the death of the placed relative, a risk factor for negative bereavement outcomes, we also expect lower levels of depression and complicated grief post-death among persons in the active treatment condition whose relative dies. In as much as the demand and utilization of long-term care is virtually certain to increase in the decades ahead, this study has the potential of providing valuable guidance in navigating this transition and in improving health outcomes for caregivers in the short- and long-term. The specific aims of this study are to:

1. Assess the effects of an intervention targeting caregivers who recently placed a relative in a long-term care facility because of cognitive and/or physical disability. In a two group randomized clinical trial we predict that caregivers assigned to active treatment will have lower levels of depressive symptoms, anxiety symptoms, and greater satisfaction with the long-term care facility when compared to individuals assigned to the control condition.
2. Assess the impact of the intervention on psychiatric outcomes and on complicated grief for those caregivers whose relative dies during follow up. We predict that long-term symptoms of depression and symptoms of complicated grief will be lower after death among caregivers assigned to active treatment when compared to those in the control condition.
3. Carry out exploratory analysis to assess the effects of the intervention on resident-related outcomes, including number of emergency room visits and hospitalizations, rate of functional decline, perceived quality of life, and formal complaints filed on behalf of the resident. Because the intervention engages the caregiver in monitoring resident health status and in end-of-life planning, we predict that resident-related outcomes will be better in the active treatment group. Overall, this should be reflected in greater perceived quality of life of residents in active treatment when compared to residents of participants in the control condition.

ELIGIBILITY:
Inclusion Criteria: The Caregiver

1. is a family member/partner (e.g., spouse, child, or fictive kin) of institutionalized person;
2. is 21 years of age or older;
3. provided a minimum of 3 months of in-home care prior to institutionalization;
4. speaks English; and
5. plans to live in the area for at least 6 months.

The care recipient/resident must:

(1) be 50 years old or older; and (2) have been permanently placed within a long-term care facility within the last 120 days with impairment in at least 3 of 6 Activities of Daily Living.

-

Exclusion Criteria:

(1) care recipient is enrolled in a hospice program.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 217 (Actual)
Dates: Start 2008-01; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Depression | 6, 12, and 18 months after baseline assessment
  Depressive affect assesed with CES-D
State Anxiety | 6, 12,and 18 months post baseline
  Assessed general anxiety using the Spielberger et al., state anxiety inventory
Caregiver Burden | 6, 12, and 18 months
  Burden as assessed by Bedard et al, adaptation of Zarit Burden interview
Complicated Grief | 6, 12, and 18 months post-baseline
  Prigerson et al, complicated grief scale; applies only to caregivers who experience the death of a loved one

SECONDARY OUTCOMES:
Prescription medication use | 6,12, and 18 months post-baseline
  Prescription medication for depression and anxiety
Social activities | 6, 12, and 18 months post-baseline
  Assesses satisfaction with time spent engagin in social activites, REACH instrument
Quality of Life AD | 6, 12, and 18 months post-baseline
  Caregivers assessment of the quality of life of AD patient using scale by Logsdon et al.,
Texas Revised Inventory of Grief | 6, 12, and 18 months post-baseline
  Fashingbauer scale used to assess grief in caregivers who experienced the death of their loved one
After-death bereaved family member interview (nursing home version) | 6, 12, and 18 months post-baseline
  Assesses resident care prior to death on four dimensions;used only for caregivers who experience the death of a loved one
Overall rating scale for patient focused, family centered care | 6, 12, and 18 months post-baseline
  Assesses overall communication, respect for patient wishes, symptom control, provided emotional support to family by nursing home staff

CONTACTS AND LOCATIONS:
Overall Officials: Richard Schulz, PH.D., Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Result] Schulz R, Rosen J, Klinger J, Musa D, Castle NG, Kane A, Lustig A. Effects of a Psychosocial Intervention on Caregivers of Recently Placed Nursing Home Residents: A Randomized Controlled Trial. Clin Gerontol. 2014 Jan 1;37(4):347-367. doi: 10.1080/07317115.2014.907594. PMID 25071302